CLINICAL TRIAL: NCT00099723
Title: The Effect of a Probiotic on Hepatic Steatosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The hypothesis that probiotics would reduce hepatic steatosis in humans was not supported
Sponsor: VSL Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SS01305-01; R21AT001305-01 (NIH)
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2004-12

CONDITIONS: Fatty Liver
Keywords: Hepatic steatosis; adult-onset diabetes; Non-alcoholic fatty liver disease
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

INTERVENTIONS:
Drug: VSL#3

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is an accumulation of fat and fibrous tissue in the liver. It is the most common cause of chronic liver disease in the United States. The exact cause of NAFLD is unknown, but it is more common among people with conditions such as adult-onset diabetes. NAFLD can strike people of all ages but most often affects adults between the ages of 40 and 60. Research indicates that overgrowth of gut bacteria can start a chain of biological processes that stress the liver, causing liver inflammation. Probiotics, living bacteria taken orally, may decrease the stress on the liver by reducing this bacterial overgrowth and/or strengthening the gut walls. Because probiotics are generally safe, inexpensive, and easy to tolerate they are an attractive treatment option for NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Adult-onset diabetes
* Liver biopsy in the previous 2 months with diagnosis of fatty liver and fibrosis stage F2-F3

Exclusion Criteria:

* There are multiple exclusion criteria.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-10; Study Completion 2005-12 (Estimated)

PRIMARY OUTCOMES:
MRI
Liver biopsy
Blood work

CONTACTS AND LOCATIONS:
Overall Officials: Steve Solga, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States